CLINICAL TRIAL: NCT04618302
Title: Test-retest Reliability of Lung Diffusing Capacity for Nitric Oxide During Light and Moderate Intensity Cycling Exercise
Brief Title: Lung Diffusing Capacity for Nitric Oxide During Cycling Exercise
Status: Completed | Type: Observational
Sponsor: Thomas Radtke (Other)
Responsible Party: Sponsor-Investigator, Thomas Radtke, PD Dr phil Thomas Radtke, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2020-01756
Record Dates: First submitted 2020-10-28; First posted 2020-11-05 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: lung diffusing capacity for nitric oxide; lung function testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the test-retest reliability of the lung diffusing capacity for nitric oxide in healthy individuals during exercise.

DETAILED DESCRIPTION:
The aim of this study of to evaluate the test-retest reliability of single-breath lung diffusing capacity measurements for nitric oxide (DLNO) in healthy individuals during light and moderate intensity cycling exercise. Healthy subjects will perform repeated single-breath DLNO measurements during light (i.e., at 50% of the first ventilatory threshold) and moderate intensity exercise (i.e., 80% of the first ventilatory threshold) on a stationary cycle ergometer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 18 yrs and older
* Ability to follow study procedures and instructions in German

Exclusion Criteria:

* Any known cardiopulmonary or metabolic diseases (e.g., heart disease, diabetes mellitus etc)
* Obesity (BMI > 30kg/m2)
* Smoking (ex-smoker allowed; if they stopped smoking at least one year before the examination)
* Mental impairment leading to inability to cooperate
* Respiratory infection in the last two weeks
* Forced expiratory volume in 1s/ forced vital capacity (FEV1/FVC ratio) FEV1/FVC ratio < lower limit of normal according to equations by Quanjer et al. Eur Respir J 2012.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy people without chronic cardiopulmonary diseases will be invited to participate in this study.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Diffusing capacity for nitric oxide (DLNO) | At second study visit
  DLNO (in ml/min/mmHg) measured at 80% of the gas exchange threshold during cycling exercise.
Diffusing capacity for nitric oxide (DLNO) | At third study visit, approximately 1-2 weeks after second study visit
  DLNO (in ml/min/mmHg) measured at 80% of the gas exchange threshold during cycling exercise.

SECONDARY OUTCOMES:
Diffusing capacity for nitric oxide (DLNO) | At second study visit
  DLNO (in ml/min/mmHg) measured at 50% of the gas exchange threshold during cycling exercise.
Diffusing capacity for nitric oxide (DLNO) | At third study visit, approximately 1-2 weeks after second study visit
  DLNO (in ml/min/mmHg) measured at 50% of the gas exchange threshold during cycling exercise.
Diffusing capacity for carbon monoxide (DLCO) | At second study visit
  DLCO (in ml/min/mmHg) measured at 50% of the gas exchange threshold during cycling exercise.
Diffusing capacity for carbon monoxide (DLCO) | At third study visit, approximately 1-2 weeks after second study visit
  DLCO (in ml/min/mmHg) measured at 50% of the gas exchange threshold during cycling exercise.
Diffusing capacity for carbon monoxide (DLCO) | At second study visit
  Agreement in DLCO (in ml/min/mmHg) measured at 80% of the gas exchange threshold during cycling exercise.
Diffusing capacity for carbon monoxide (DLCO) | At third study visit, approximately 1-2 weeks after second study visit
  Agreement in DLCO (in ml/min/mmHg) measured at 80% of the gas exchange threshold during cycling exercise.
Alveolar volume (VA) | At second study visit
  VA (in L) measured at 50% of the gas exchange threshold during cycling exercise.
Alveolar volume (VA) | At third study visit, approximately 1-2 weeks after second study visit
  VA (in L) measured at 50% of the gas exchange threshold during cycling exercise.
Alveolar volume (VA) | At second study visit
  Alveolar volume (in L) measured at 80% of the gas exchange threshold during cycling exercise.
Alveolar volume (VA) | At third study visit, approximately 1-2 weeks after second study visit
  Alveolar volume (in L) measured at 80% of the gas exchange threshold during cycling exercise.
Breath hold time (BHT) | At second study visit
  BHT (in s) measured at 80% of the gas exchange threshold during cycling exercise.
Breath hold time (BHT) | At third study visit, approximately 1-2 weeks after second study visit
  BHT (in s) measured at 80% of the gas exchange threshold during cycling exercise.
Breath hold time (BHT) | At second study visit
  BHT (in s) measured at 50% of the gas exchange threshold during cycling exercise.
Breath hold time (BHT) | At third study visit, approximately 1-2 weeks after second study visit
  BHT (in s) measured at 50% of the gas exchange threshold during cycling exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Radtke, PhD, Principal Investigator — University of Zurich and University Hospital Zurich
Locations (1):
- University of Zurich and University Hospital of Zurich, Zurich, Switzerland